CLINICAL TRIAL: NCT00444223
Title: The Biodistribution of N-{4-[3'-[F-18] Fluoroethylphenyl)Amino]-6-quinazolinyl}-Acrylamide ([F-F18]FEQA) in Patients With Advanced Non-Small-Cell Lung Cancer (NSCLC) and in Healthy Subjects: A Pilot Study
Brief Title: Fluorine F 18 FEQA in Patients With Stage III or Stage IV Non-Small Cell Lung Cancer and in Healthy Participants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000529363; UCLA-0304039-01
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fluorine F 18 FEQA + positron emission tomography (Experimental)
  Interventions: Procedure: fluorine F 18 FEQA + positron emission tomography

INTERVENTIONS:
Procedure: fluorine F 18 FEQA + positron emission tomography

SUMMARY:
RATIONALE: Fluorine F 18 FEQA may be an effective radioactive drug to use with positron emission tomography (PET) scans.

PURPOSE: This clinical trial is studying the use of fluorine F 18 FEQA in patients with stage III or stage IV non-small cell lung cancer and in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the biodistribution of fluorine F 18 FEQA in patients with stage III or IV non-small cell lung cancer (NSCLC) and in healthy participants.
* Determine whether fluorine F 18 FEQA can be used as an imaging agent with positron emission tomography in patients with stage III or IV NSCLC.

OUTLINE: This is a pilot study.

Patients and healthy participants receive fluorine F 18 FEQA IV and then undergo whole-body dynamic scans comprising positron emission tomography.

Blood is collected during and after imaging to measure radioactivity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Must meet 1 of the following criteria:
* Diagnosis of non-small cell lung cancer by CT scan, bone scan, or biopsy

  * Stage III or IV disease
  * Clinically assessed with
* Healthy participant

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-05-04 (Actual); Primary Completion 2008-05-15 (Actual); Study Completion 2008-05-15 (Actual)

PRIMARY OUTCOMES:
Biodistribution of fluorine F 18 FEQA | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States